CLINICAL TRIAL: NCT07323979
Title: The Effects of Different Prone Positioning Angles on Cardiopulmonary Function in Children After Congenital Heart Disease Surgery: A Randomized Controlled Trial
Acronym: PACE-CHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY-Z-2022-311-04; KD022024023 (Other Grant/Funding Number: Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences))
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: CHD; Heart Defects, Congenital; Hypoxia; Respiratory Insufficiency; Postoperative Complications
MeSH Terms: conditions — Heart Defects, Congenital; Hypoxia; Respiratory Insufficiency; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: people processing the numbers (statisticians) and recording the numbers (data collectors)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10° Head-Elevated Prone Position (Experimental): Participants assigned to this group receive prone positioning therapy with the head of the bed elevated to an angle of 10 degrees. The angle is calibrated using a protractor. The prone position is maintained for at least 12 hours per day.
  Interventions: Procedure: 10° Head-Elevated Prone Positioning
- 30° Head-Elevated Prone Position (Experimental): Participants assigned to this group receive prone positioning therapy with the head of the bed elevated to an angle of 30 degrees. The angle is calibrated using a protractor. The prone position is maintained for at least 12 hours per day.
  Interventions: Procedure: 30° Head-Elevated Prone Positioning
- 45° Head-Elevated Prone Position (Experimental): Participants assigned to this group receive prone positioning therapy with the head of the bed elevated to an angle of 45 degrees. The angle is calibrated using a protractor. The prone position is maintained for at least 12 hours per day.
  Interventions: Procedure: 45° Head-Elevated Prone Positioning

INTERVENTIONS:
Procedure: 10° Head-Elevated Prone Positioning — Participants receive prone positioning therapy with the head of the bed elevated strictly to 10 degrees, verified by a protractor. The position is maintained for at least 12 hours daily. The head position is alternated every 2 hours, and arms are placed alongside the torso.
  Arms: 10° Head-Elevated Prone Position
Procedure: 30° Head-Elevated Prone Positioning — Participants receive prone positioning therapy with the head of the bed elevated strictly to 30 degrees, verified by a protractor. The position is maintained for at least 12 hours daily. The head position is alternated every 2 hours, and arms are placed alongside the torso.
  Arms: 30° Head-Elevated Prone Position
Procedure: 45° Head-Elevated Prone Positioning — Participants receive prone positioning therapy with the head of the bed elevated strictly to 45 degrees, verified by a protractor. The position is maintained for at least 12 hours daily. The head position is alternated every 2 hours, and arms are placed alongside the torso.
  Arms: 45° Head-Elevated Prone Position

SUMMARY:
The goal of this randomized controlled trial is to learn if different head-elevated prone positioning angles can optimize cardiopulmonary function and enteral nutrition tolerance in infants and children after congenital heart disease (CHD) surgery. The main questions it aims to answer are:

1. Do specific prone positioning angles (10°, 30°, or 45°) lead to better improvements in cardiopulmonary recovery, specifically regarding oxygenation, lung compliance, airway resistance, and hemodynamic stability?
2. Does increasing the elevation angle improve the tolerance of enteral nutrition (tube feeding) while maintaining patient safety?

Researchers will compare three different head-of-bed elevation angles (10°, 30°, and 45°) to see if a specific angle offers superior heart and lung support and nutritional benefits during the early postoperative period.

Participants will:

1. Be randomly assigned to one of three groups: 10°, 30°, or 45° head-elevated prone position.
2. Maintain the assigned prone position for at least 12 hours daily.
3. Undergo monitoring of cardiopulmonary indicators (including oxygen levels, ventilator parameters, blood pressure, and central venous pressure) and digestive function (gastric residual volume) at scheduled intervals (0, 4, 6, and 12 hours).

ELIGIBILITY:
Inclusion Criteria:

* Congenital Heart Disease (CHD) confirmed by echocardiography with surgery performed.

RACHS-1 score ≥ 2.

Postoperative acute hypoxemia, defined as PaO2/FiO2 ≤ 100 mmHg with bilateral infiltrates.

Receiving invasive mechanical ventilation.

Nasogastric or nasoenteric tube in place.

Hemodynamic stability for ≥ 72 hours (inotropic score ≤ 25).

Exclusion Criteria:

* Cardiac arrest or age-specific bradycardia (> 20% below normal).

Active bleeding.

Significant pneumothorax.

Delayed sternal closure.

Transfer to another facility or death before completing the protocol.

Withdrawal of consent by legal guardians.

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Lung Compliance | Baseline (0 hours), 4 hours, and 6 hours after initiation of prone positioning.
Oxygenation Index (OI) | Baseline (0 hours), 4 hours, and 6 hours after initiation of prone positioning.
  The Oxygenation Index is a measure used to assess the severity of hypoxic respiratory failure and lung function recovery. It is calculated using the formula: OI = (FiO2 × Mean Airway Pressure × 100) / PaO2. Arterial blood gases (PaO2) are obtained from arterial lines, and FiO2 and mean airway pressure are recorded from the ventilator. Lower scores indicate better oxygenation status.
Airway Resistance | Baseline (0 hours), 4 hours, and 6 hours after initiation of prone positioning.
  Airway resistance is measured by the mechanical ventilator to assess the resistance of the respiratory tract to airflow. Lower values indicate better airway patency and less obstruction. Unit: cmH2O/L/s.

SECONDARY OUTCOMES:
Gastric Residual Volume (GRV) | Baseline (0 hours), 6 hours, and 12 hours after initiation of prone positioning.
  Gastric residual volume is assessed by aspirating gastric contents through the nasogastric tube before feeding. It serves as a key indicator of enteral nutrition tolerance and gastric emptying function. Lower volumes indicate better tolerance and faster gastric emptying. Unit: mL.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Privacy confidentiality